CLINICAL TRIAL: NCT04107987
Title: An Evaluation of a Nutraceutical With Berberine, Curcumin, Inositol, Banaba and Chromium Picolinate in Patients With Fasting Dysglycemia
Brief Title: Berberine, Curcumin, Inositol, Banaba and Chromium Picolinate in Patients With Fasting Dysglycemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, MD, PHd, FESC, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P-20180017962
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Dysglycemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reglicemi (Active Comparator): Reglicemi is a nutraceutical containing Berberine, Curcumin, Inositol, Banaba, and Chromium Picolinate
  Interventions: Dietary Supplement: Reglicem
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Reglicem — Reglicem is a nutraceutical containing Berberine, Curcumin, Inositol, Banaba, and Chromium Picolinate
  Arms: Reglicemi
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Dysglycemia is an important pre-risk condition which can potentially lead to diabetes if not adequately treated. The variation of glycemic balance can lead to cardiovascular disorders. The study will evaluate if Reglicem®, a nutraceutical containing Berberine, Curcumin, Inositol, Banaba, and Chromium Picolinate, can ameliorate glycemic status in patients with dysglycemia.

DETAILED DESCRIPTION:
Dysglycemia is an important pre-risk condition which can potentially lead to diabetes if not adequately treated. The variation of glycemic balance can lead to cardiovascular disorders. The study will evaluate if Reglicem®, a nutraceutical containing Berberine, Curcumin, Inositol, Banaba, and Chromium Picolinate, can ameliorate glycemic status in patients with dysglycemia.

The investigators will enroll patients with impaired fasting glucose (IFG) or impaired glucose tolerance (IGT), not taking other hypoglycemic compounds. Patients will be randomized to take Reglicem® or placebo for 3 months, in a randomized, double-blind, placebo-controlled design. Reglicem® and placebo will be self-administered once a day, 1 tablet during the breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Patients with impaired fasting glucose (IFG) or impaired fasting glucose (IGT)
* Patients not taking hypoglycemic agents (both pharmaceuticals or nutraceutical agents)

Exclusion Criteria:

* Patients with type 1 or type 2 diabetes mellitus
* Patients with impaired hepatic function
* Patient with impaired renal function
* Patients with gastrointestinal disorders
* Patients with current or previous evidence of ischemic heart disease, heart failure, or stroke
* Patients with weight change of > 3 Kg during the preceding 3 months
* Patients with hystory of malignancy, and significant neurological or psychiatric disturbances, including alcohol or drug abuse.
* Patients taking (within the previous 3 months) hypoglycemic agents, laxatives, beta-agonists (other than inhalers), cyproheptadine, anti-depressants, antiserotoninergics, phenothiazines, barbiturates, oral corticosteroids, and antipsychotics
* Women who were pregnant or breastfeeding or of childbearing potential and not taking adequate contraceptive precautions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Progression of dysglicemia | 3 months
  Oral glucose tolerance test

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Matteo, Pavia, Lombardy, Italy